CLINICAL TRIAL: NCT05946395
Title: Comparison of Synchronous or Delayed Speech Therapy and Audioprosthetic Care in Older Adults With First-time Hearing Aids
Brief Title: Comparison of Speech Therapy and Audioprosthetic Care in Older Adults With First-time Hearing Aids
Acronym: CODITION
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor, in consultation with the coordinating investigator, decided to stop the study prematurely on 23/10/2024. Unfortunately, no patients were included in the study.
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A02788-35
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided by drawing lots into 2 groups. Group A will benefit from speech therapy and synchronous equipment, and group B will begin speech therapy after 3 months after the installation of the equipment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing aid and synchronous speech therapy (Experimental): This arm will begin speech therapy at the same time as the fitting of the hearing aid.
  Interventions: Device: Hearing aid; Other: Speech therapy session
- Hearing aid and deferred speech therapy (Active Comparator): This arm will begin speech therapy 3 months after fitting the device.
  Interventions: Device: Hearing aid; Other: Speech therapy session

INTERVENTIONS:
Device: Hearing aid — Fitting a hearing aid
Other: Speech therapy session — As speech therapy is part of standard care, the objective of the study will be to compare the impact of synchronous or delayed audioprosthetic and speech therapy care on the impact of deafness in elderly patients.

SUMMARY:
The purpose of the study is to evaluate the score of the Evaluation of the Impact of Deafness in Adults(ERSA)/150 questionnaire obtained at 3 months compared to the inclusion score.

DETAILED DESCRIPTION:
This is a pilot, prospective, interventional, comparative, randomized, longitudinal, open, multicenter study comparing synchronous and delayed hearing aid and speech therapy.

Patients will be randomly divided by drawing lots into 2 groups. Both groups will benefit from a hearing aid prescription and speech therapy for a series of 24 sessions at the rate of 1 per week, for an approximate duration of 6 months. Group A will benefit from speech therapy and synchronous equipment, and group B will begin speech therapy after 3 months after the installation of the equipment.

Regarding the equipment, it will not be the same for all patients. Indeed, it is the one that will best suit the patient who will be chosen. The same will apply to the settings, in accordance with the usual support.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 65 to 80;
* First equipment;
* Average hearing loss between 40 and 70 db;
* Speech comprehension greater than 50%;
* Absence of acoustic recruitment phenomenon;
* Symmetrical bilateral deafness (inter aural difference <20dB);
* Affiliated patient or beneficiary of a social security scheme;
* Patient speaking and understanding French, able to complete questionnaires and scales;
* Patient having been informed and having signed an informed consent to participate in the study.

Exclusion Criteria:

* Patient with a psychiatric pathology;
* Patient with neurological disorders;
* Patient taking psychotropic drugs;
* Patient participating in another clinical study;
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision;
* Patient hospitalized without consent.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Impact of Deafness in Adults | 3 months
  Score of the questionnaire "Assessment of the Impact of Deafness in Adults" obtained at 3 months compared to the inclusion score.
  The ERSA (Evaluation of the Repercussions of Deafness in Adults) assesses four areas: quality of life, personal life, social life and professional life. It is rated out of 200 or out of 150 in the absence of professional life. The higher the ERSA score, the better the patient's quality of life.

IPD SHARING:
Plan to Share IPD: No